CLINICAL TRIAL: NCT04335448
Title: Comprehensive Long-term Follow up of Adults With Arterial Switch Operation - European Collaboration for Prospective Outcome Research in Congenital Heart Disease
Brief Title: Comprehensive Long-term Follow up of Adults With Arterial Switch Operation
Acronym: EPOCH-ASO
Status: Active, not recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Matthias Greutmann, PD. Dr. med., University of Zurich
Other Study IDs: EPOCH
Record Dates: First submitted 2020-03-23; First posted 2020-04-06 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Transposition of Great Vessels
Keywords: transposition of the great arteries; arterial switch operation; coronary artery anomaly; outcome
MeSH Terms: conditions — Transposition of Great Vessels

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Arterial Switch Operation - Transposition of Great Arteries: Patients with previous arterial switch operation for the treatment of a transposition of great arteries will constitute the sole group of the cohort.
  Interventions: Other: No intervention is planed

INTERVENTIONS:
Other: No intervention is planed — No intervention is planed

SUMMARY:
Background: Long-term outcomes in adults with prior arterial switch operation (ASO) have not yet been well defined. The aim of this study is to elucidate incidence and predictors of adverse cardiac outcomes in a prospectively followed cohort of adults after their ASO.

Methods: The comprehensive long-term follow up of adults with ASO is a project within the European collaboration for prospective outcome research in congenital heart disease (EPOCH). It is designed as a prospective, international multicenter cohort study. Consecutive patients (aged 16 years or more) with prior ASO will be included at 11 European tertiary care centers. Participants will be followed according to a standardized protocol following international recommendations, including standardized protocols for imaging and for exercise testing. Main outcome measures are all-cause and cardiac-related mortality, rate of cardiac re-intervention, neo-aortic dissection, myocardial infarction, stroke, infective endocarditis, sustained atrial and ventricular arrhythmias, new-onset or worsening pulmonary hypertension and new-onset heart failure. Secondary endpoints are frequency and progression of right ventricular outflow tract stenosis, neo-aortic root dilatation, neo-aortic valve regurgitation and ventricular dysfunction. The impact of demographic, anatomic (e.g. coronary artery anatomy) and functional variables on the above-mentioned outcomes, as well as quality of life and incidence of pregnancy related complications will also be assessed.

Aim: The prospective, international, multicenter EPOCH-ASO study will provide a better understanding of adverse outcomes and their predictors in adults after ASO. The results of the EPOCH-ASO study may help to optimize future care of this novel patient cohort in adult cardiology.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥16 years)
* with transposition of great arteries or a Taussig-Bing anomaly
* who underwent repair by an ASO, and who are actively followed at one of the participating centers will be enrolled.

Exclusion Criteria:

* Incapability of giving informed consent and previous heart transplant.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adults (≥16 years) with transposition of great arteries or a Taussig-Bing anomaly who underwent repair by an ASO, and who are actively followed at one of the participating centers will be enrolled. Exclusion criteria are incapability of giving informed consent and previous heart transplant.
Sampling Method: Non-Probability Sample
Enrollment: 540 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2039-09-30 (Estimated); Study Completion 2039-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of all-cause mortality | during a follow up of up to 20 years
  Determination of cause of death
Incidence of cardiac-related mortality | during a follow up of up to 20 years
  Sudden cardiac death (death that ensues unexpected within one hour of onset of symptoms), death related to acute myocardial infarction, death that is primarily caused by heart failure or death within 30 days or during the hospital admission after a cardiac intervention.
Incidence/rate of re-intervention | during a follow up of up to 20 years
  Includes all types of cardiac re-intervention with detailed analysis of the indication of re-intervention.
Incidence/rate of neo-aortic dissection | during a follow up of up to 20 years
  Aortic dissection with entry within the neo-aortic root.
Incidence of myocardial infarction | during a follow up of up to 20 years
  Defined according to the Fourth Universal Definition of Myocardial Infarction. Defined according to the Fourth Universal Definition of Myocardial Infarction.
Incidence of arrhythmias | during a follow up of up to 20 years
  Atrial arrhythmias with a duration of >30 seconds, or requiring anti-arrhythmic medication or ablation procedures and / or sustained ventricular tachycardia (heart rate >100/min) for at least 30 seconds or requiring electrical cardioversion / defibrillation.
Incidence of new onset / worsening heart failure | during a follow up of up to 20 years
  Hospital admission for heart failure or initiation of heart failure medication for symptoms of heart failure (excludes initiation of medication for asymptomatic deterioration of ventricular function), according to the current guidelines of the European Society of Cardiology.
Incidence of stroke | during a follow up of up to 20 years
  Focal neurological symptoms and confirmation of cerebral ischemia or infarction by cerebral magnetic resonance imaging or computed tomography.
Incidence of infective endocarditis | during a follow up of up to 20 years
  Defined according to the modified Duke's criteria, according to the current ESC guidelines.
Incidence of pulmonary hypertension | during a follow up of up to 20 years
  Defined as an increase in mean pulmonary arterial pressure (PAPm) ≥20 mmHg at rest as assessed by right heart catheterization.

SECONDARY OUTCOMES:
Rate of right ventricular outflow tract stenosis | during a follow up of up to 20 years
  At least 1 of the following criteria:
  * Branch pulmonary artery minimal diameter: maximal diameter at least 1:2 on CT or MRI
  * Echocardiographic systolic peak gradient across branch pulmonary arteries > 16mmHg (peak velocity > 2.0m/s)
  * Estimated right ventricular systolic pressure > 40mmHg (determined by RV/RA-pressure gradient and estimated central venous pressure, see echocardiography protocol for details)
Rate of the different patterns of the coronary anatomy | during a follow up of up to 20 years
  To study the impact of coronary artery anatomy and type of coronary reimplantation on cardiovascular morbidity, ventricular function and functional capacity with a specific focus on presence of coronary artery obstruction, acute proximal angulation and inter-arterial or intramural course.
Incidence/rate of neo-aortic root dilatation | during a follow up of up to 20 years
  Increase of neo-aortic root dilatation of at least 3mm, determined with the same imaging modality and appropriate side-by-side comparison of actual images.
Incidence of progression of neo-aortic root dilatation | during a follow up of up to 20 years
  Increase of neo-aortic root dilatation of at least 3mm, determined with the same imaging modality and appropriate side-by-side comparison of actual images.
Incidence/rate of neo-aortic regurgitation | during a follow up of up to 20 years
  Assessment by echocardiography:
  - Mild, moderate, severe (50)
  Assessment by CMR
  - Regurgitation fraction and volume by flow measurements in proximal aortic root.
Incidence of progression of neo-aortic regurgitation | during a follow up of up to 20 years
  Increase > 1 grade (echocardiography) Increase of regurgitant fraction >10% on CMR.
Incidence/rate of left ventricular systolic dysfunction | during a follow up of up to 20 years
  Echocardiography:
  - Left ventricular ejection fraction (LVEF) biplane Simpson <52% for men and <54% for women (33)
  CMR:
  - LVEF < 52%
Incidence/rate of left ventricular diastolic dysfunction | during a follow up of up to 20 years
  Echocardiography:
  - Defined according to the current recommendations for the evaluation of left ventricular diastolic function by the America society of echocardiography and the European association of cardiovascular Imaging.
Incidence of worsening left ventricular function | during a follow up of up to 20 years
  Decrease of LVEF >5%
Incidence/rate of Right ventricular dysfunction | during a follow up of up to 20 years
  Echocardiography:
  - At least 2 of the following
  * FAC <30%
  * TAPSE <18mm
  * TAPSE S' <10cm/s
  CMR:
  - RVEF < 50%
Incidence of worsening right ventricular function | during a follow up of up to 20 years
  Echocardiography (not valid in case of worsening tricuspid regurgitation) - At least 2 of the following:
  * Decrease in Fac > 10%
  * Decrease in TAPSE >5mm
  * Decrease in TAPSE S' >3cm/s
  CMR:
  - Decrease in RVEF >5%
Rate of poor functional capacity | during a follow up of up to 20 years
  As determined by cardiopulmonary exercise testing by measuring Lung Function (flow volume loops), oxygen consumption during exercise (VO2 max), anaerobic threshold, heart performance during exercise (O2-Heart rate)
Incidence of pregnancy | during a follow up of up to 20 years
  To study the impact of pregnancy on mortality and cardiovascular morbidity.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Greutmann, MD, Principal Investigator — University of Zurich
Locations (11):
- University Hospital Vienna, Vienna, Austria
- CHU Paris IdF Ouest - HEGP Hôpital Européen Georges Pompidou, Paris, France
- Amsterdam University Medical Center, Amsterdam, Netherlands
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario y Politécnico La Fe Valencia, Valencia
- Switzerland (5):
  - University Hospital Basel, Basel
  - University Hospital Inselspital Bern, Bern
  - University Hospital Geneva, Geneva
  - University Hospital Lausanne, Lausanne
  - University Hospital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ruperti-Repilado FJ, Ladron R, Lopez-Ayala P, Gabra B, Gonzalez-Fernandez V, Engele LJ, Manso B, Bouma BJ, Gabriel H, Schwitz F, Possner M, Schwerzmann M, Rueda J, Buendia-Fuentes F, Bouchardy J, Ladouceur M, Dos-Subira L, Greutmann M, Tobler D, Gallego P. Aortic coarctation and long-term morbidity after arterial switch operation: a multicentre international cohort study. Heart. 2025 Jul 23:heartjnl-2024-325634. doi: 10.1136/heartjnl-2024-325634. Online ahead of print. PMID 40701798

DOCUMENTS (1):
  • Study Protocol (2019-08-24): https://cdn.clinicaltrials.gov/large-docs/48/NCT04335448/Prot_000.pdf